CLINICAL TRIAL: NCT03273621
Title: Effetti di Differenti Tipologie di Intervento di Chirurgia Bariatrica Sul Tessuto Adiposo Epicardico e su Alcuni Parametri Morfologici e Funzionali Cardiovascolari, Valutati Con Risonanza Magnetica Nucleare
Brief Title: Bariatric Surgery and Epicardial Adipose Tissue: a MRI Study
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Head of Radiology Department, IRCCS Policlinico S. Donato
Other Study IDs: EAT-BS _01
Record Dates: First submitted 2017-07-10; First posted 2017-09-06 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese: Patients with a body mass index larger than 35 kg/m2
  Interventions: Procedure: Bariatic surgery

INTERVENTIONS:
Procedure: Bariatic surgery — One of two different types of surgery: sleeve gastrectomy and Roux-en-Y gastric by-pass.

SUMMARY:
The aim of this study is to measure the volume of the epicardial adispose tissue (EAT) and other morphological and functional cardiovascular parameters in subjects with severe obesity, using an open magnetic resonance unit capable of holding up to 220 kg of weight. These measurements will be repeated a year after bariatric surgery to assess the effect of the weight loss on EAT. The possible difference among different types of bariatric surgery will be considered.

DETAILED DESCRIPTION:
In this prospective observational study, 28 obese male and female subjects underwent bariatric surgery will be studied: 14 subjects candidates for SG and 14 at RYGB. These patients will enrolled in this type of intervention at the INCO bariatric surgery unit (National Institute for Obesity). All patients are first evaluated by a multidisciplinary team to establish adherence to the criteria suggested by the guidelines for bariatric surgery.

All enrolled subjects will be subjected to the following protocol within one month prior to surgery and one year (±1 month) after surgery:

1. CMR without contrast medium with 1-T (Panorama, Philips) open device for the measurement of EAT volume in systoles and diastoles for the evaluation of the main morpho-functional parameters (left ventricular size and mass , Right ventricular size, atrial size, left and right ventricular systolic function, diastolic left and right ventricular function) and for evaluating the elasticity of the thoracic aortic wall, evaluated as compliance and stiffness (duration of examination About 30 minutes).
2. performing axial MRI scans without contrast medium at the IV lumbar vertebra for quantification of abdominal and subcutaneous adipose tissue;
3. direct detection of anthropometric indexes (weight, height, abdominal circumference, hip circumference);
4. measurement of systolic and diastolic blood pressure with sphygmomanometer;
5. assessment of body composition by bioimpedenzometry with estimate of fat and lean mass expressed in kg and in percentage.

The examinations will be carried out following the normal procedures provided by clinical practice and all scans performed by Magnetic Resonance will be performed at the Italian Diagnostic Center (CDI), Via Saint Bon, 20 - 20147 Milan (which has MRI equipment open). Other investigations will be carried out at the Istituto Nazionale per la cura del dono (INCO) of the Sant'Ambrogio Clinical Institute.

The sample size was calculated assuming that an average thickness of 12.3±1.8 mm (Iacobellis G. at al, 2008) is expected to reduce the thickness by approximately 30% to 4 ± 0.8 mm (from An average epicardial fat content of 137 ± 37 ml is expected to be about 30% reduction of 39 ± 12 ml). With a 90% power and alpha error of 5% (two-tailed) we have obtained a minimum number of 22 subjects. Assuming a 20% loss to follow-up, approximately 28 subjects should be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. patients with bariatric surgery
2. informed written consent
3. between the ages of 18 and 65
4. patients with body mass index (BMI) ≥ 40 kg / m2
5. patients with 35 ≤ BMI <40 kg / m2 in the presence of comorbidities that could improve or cure following the remarkable and persistent weight loss achieved with the intervention (metabolic diseases, cardiorespiratory diseases, severe joint disorders, severe psychological problems, etc.)
6. patients with 35 ≤ BMI <40 kg / m2 with previous failure of proper medical treatment (lack or insufficient weight loss, lack or lack of long-term maintenance of weight loss).

Exclusion Criteria:

1. lack of informed written consent
2. presence of known ischemic or valvular heart disease
3. pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
EAT volume | Immediately after MRI
  The EAT volume will be measured in ml by manul segmentation of magnetic resonance images
EAT thickness | Immediately after MRI
  The EAT maximal thickness will be measured in mm by using an electronic caliper on magnetic resonance images

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica San'Ambrogio, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided